CLINICAL TRIAL: NCT07379658
Title: Improving HIV Prevention Outcomes: Insights on Long-Acting Injectable (LAI) HIV Pre-Exposure Prophylaxis (PrEP) Patient-Reported Medication Preferences, Adherence, and Clinical Outcomes (IMPACT) in a Southern US State
Brief Title: Long-Acting Injectable HIV PrEP PROs
Acronym: IMPACT
Status: Not yet recruiting | Type: Observational
Sponsor: Anupama Raghuram MD (Other)
Collaborators: Gilead Sciences (Industry); University of Louisville (Other)
Responsible Party: Sponsor-Investigator, Anupama Raghuram MD, Chief Research Scientist, Norton Healthcare
Organization: Norton Healthcare (Other)
Other Study IDs: 25-N0026
Record Dates: First submitted 2026-01-05; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: HIV Pre-exposure Prophylaxis
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- LEN LAI PrEP: Those receiving or initiating LEN LAI PrEP
  Interventions: Other: Interview and survey to evaluate patient reported outcomes between the two medications.
- CAP LAI PrEP: Those receiving or initiating CAB LAI PrEP
  Interventions: Other: Interview and survey to evaluate patient reported outcomes between the two medications.

INTERVENTIONS:
Other: Interview and survey to evaluate patient reported outcomes between the two medications. — No intervention, the two cohorts will receive the same surveys and interviews.

SUMMARY:
The goal of this observational study is to learn about the real world effectiveness, patient satisfaction and clinical outcomes of LAI PrEP with lenacapavir (LEN) versus cabotegravir (CAB) through surveys and interviews.

Participants receiving or initiating LAI PrEP part of their regular medical care will complete surveys and interviews at three study visits over the course of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 and older
2. Deemed eligible for HIV PrEP per healthcare provider
3. Receiving or initiating LAI PrEP, defined as:

   1. Current use of CAB or LEN LAI PrEP at study entry
   2. Initiation of either CAB or LEN LAI PrEP within 30 days of study enrollment
4. Receiving PrEP services in Louisville, KY
5. Able to provide informed consent and complete study assessments

Exclusion Criteria:

1. HIV diagnosis prior to enrollment
2. Currently on oral PrEP with no plans to switch to LAI PrEP
3. Hypersensitivities to LEN or CAB
4. Pregnant or planning to become pregnant
5. PI discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving injectable PrEP in Louisville, KY.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
LAI-SQ-6 Survey, Long-Acting Injectable Satisfaction Questionnaire | Time of Enrollment, 6 months, 12 months
  The primary endpoint of this study is to compare treatment satisfaction of CAB and LEN LAI PrEP, as measured by the Long-Acting Injectable Satisfaction Questionnaire (LAI-SQ-6), adapted for LAI therapy from the Treatment Satisfaction Questionnaire for Medication- 9 (TSQM-9) [12]. The minimum score possible on this questionnaire is 0 and the maximum score possible on this questionnaire is 36. Higher scores indicate a higher satisfaction, while lower scores suggest areas for improvement in patient experience with injectable medication.

SECONDARY OUTCOMES:
Persistence with Injectable PrEP | 6 months and 12 months
  Calculated by the proportion of days covered (PDC) and identification of gaps in treatment using medication administration data.
Injection Adherence | Enrollment, 6 months, 12 months
  Measured by the Injection Adherence Rating Scale (IARS). The IARS is a Yes/No questionnaire intended to capture valuable insight from patients using long-acting injectable medications, allowing providers to improve adherence by addressing concerns related to adherence to injection schedule, perception of the injection, and the impact of side effects. .
  A patient is considered adherent if they answer "No" to questions 1-5 and "Yes" to questions 7-8 (indicating consistent attendance to injections, confidence in the protective effect of the medication, and positive engagement with the regimen).
  A patient is considered non-adherent if they answer "Yes" to questions 1-5 (indicating missed or delayed injections due to forgetfulness or lack of consistency) or "Yes" to questions 9-10 (indicating negative feelings about the injection process, which may signal discomfort or side effects affecting adherence).
Injection Site Reactions | Enrollment, 6 months, 12 months
  Injection Site Reaction Questionnaire (ISRQ) for patient-reported symptoms - DAIDS criteria for grading of infusion and injection site reactions. The ISRQ is a Yes/No questionnaire and is a tool intended to capture valuable insight from patients using long-acting injectable medications, allowing providers to assess patient perceived severity of reactions to injectable drugs.
  Scoring and Interpretation:
  Mild Injection Site Reaction (ISR): A patient is considered to have mild ISR if they respond "Yes" to 1-2 symptoms.
  Moderate ISR: A patient is considered to have moderate ISR if they respond "Yes" to 3 symptoms.
  Severe ISR: A patient is considered to have severe ISR if they respond "Yes" to ≥ 4 symptoms.
HIV Prevention Effectiveness | Baseline, 6 months, and 12 months
  Reviewing HIV test results to confirm new HIV diagnoses during the study period.
Incidence of Co-occurring STIs | Enrollment, 6 months, and 12 months
  Reviewing routine STI testing outcomes to determine the incidence of Co-occurring STIs.
Patient perceptions and preferences | Enrollment, 6 months, and 12 months
  Explored in a subset of 20 patients through the injectable PrEP Experience Interview (IPEI).
Retention in Care | 6 months and 12 months
  Evaluated through the proportion of appointments attended (PAA) and the proportion of patients with a scheduled end-of-study visit (PESV).
Visit Burden Index | 6 months and 12 months
  Evaluated through the number of PrEP-related visits per patient (i.e. provider visits, injection visits, laboratory visits, and urgent/ emergency department visits for adverse reactions to PrEP and/or additional STI screening).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Norton Healthcare, Louisville, Kentucky
  - University of Louisville, School of Public Health and Information Sciences, Louisville, Kentucky
  - University of Louisville, Kent School of Social Work, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS. Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse, Corrected version 2.1. [July 2017]. Available from https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf
- [Background] Lee, E., et al(2010). PMS36 Injection Site Reaction Questionnaire: An Adequate Tool For Measuring Injection Site Reactions? Value in Health, 13(3), A129.
- [Background] Thompson, K, et al. Reliability and validity of a new Medication Adherence Rating Scale (MARS) for the psychoses. Schizophrenia research. 42. 241-7. 10.1016/S0920-9964(99)00130-9.
- [Background] Bharmal M, et al. Validation of an abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9) among patients on antihypertensive medications. Health Qual Life Outcomes. 2009;7:36.
- [Background] Woodcock A, Bradley C. Validation of the revised 10-item HIV Treatment Satisfaction Questionnaire status version and new change version. Value Health. 2006 Sep-Oct;9(5):320-33. doi: 10.1111/j.1524-4733.2006.00121.x. PMID 16961550
- [Background] Kelley CF, et al.Twice-Yearly Lenacapavir for HIV Prevention in Men and Gender-Diverse Persons. N Engl J Med. 2024 Nov 27. 10. Murray MI, et al. Satisfaction and acceptability of cabotegravir long-acting injectable suspension for prevention of HIV: Patient perspectives from the ECLAIR trial. HIV Clin Trials. 2018;19(4):129-138.
- [Background] Bekker LG, et al. Twice-Yearly Lenacapavir or Daily F/TAF for HIV Prevention in Cisgender Women. N Engl J Med. 2024 Oct 3;391(13):1179-1192.
- [Background] Hojilla JC, et al. Characterization of HIV Preexposure Prophylaxis Use Behaviors and HIV Incidence Among US Adults in an Integrated Health Care System. JAMA Netw Open. 2021;4(8):e2122692.
- [Background] Nunn AS, et al. Defining the HIV pre-exposure prophylaxis care continuum. Aids. 2017 Mar 13;31(5):731-4.
- [Background] CDC. Core indicators for monitoring the Ending the HIV Epidemic initiative: National HIV Surveillance System data reported through September 2023; and PrEP data reported through June 2023. https://www.cdc.gov/hiv/library/reports/surveillance-data-tables. Published December 2023. Accessed March 28, 2025.
- [Background] Singh, S., et al. Estimating Lifetime Risk of a Diagnosis of HIV Infection Among MSM: United States, 2017-2021. Conference on Retroviruses and Opportunistic Infections, Denver, Colorado, March 3-6 2024 https://www.natap.org/2024/CROI/croi_243.htm
- [Background] HIV/AIDS Reporting and Statistics - Cabinet for Health and Family Services. HIV/AIDS Annual Surveillance Report 2024. Ky.gov. https://www.chfs.ky.gov/agencies/dph/dehp/hab/Pages/reportsstats.aspx, accessed March 14, 2025
- [Background] Centers for Disease Control and Prevention. (2024, April 22). Fast Facts: HIV in the United States. CDC.gov. https://www.cdc.gov/hiv/data-research/facts-stats/index.html, accessed March 14, 2025
- [Background] CDC. (2024). Expanding PrEP Coverage in the United States to Achieve EHE Goals. National Center for HIV, Viral Hepatitis, STD, and Tuberculosis Prevention. https://www.cdc.gov/nchhstp/director-letters/expanding-prep-coverage.html, accessed March 14, 2025